CLINICAL TRIAL: NCT00000829
Title: A Double-Blind Placebo-Controlled Trial of the Safety and Immunogenicity of a Seven Valent Pneumococcal Conjugate Vaccine in Presumed HIV-Infected Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Lederle-Praxis Biologicals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACTG 292; 11268 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pneumococcal Infections
Keywords: Vaccines, Synthetic; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Pneumococcal Infections; Bacterial Vaccines
MeSH Terms: conditions — HIV Infections; Pneumococcal Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Patients receiving intramuscular heptavalent pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal Vaccine, Polyvalent (23-valent); Biological: Pneumococcal Conjugate Vaccine, Heptavalent
- 2 (Placebo Comparator): Patients receiving placebo vaccine
  Interventions: Biological: Pneumococcal Vaccine, Polyvalent (23-valent); Biological: Placebo

INTERVENTIONS:
Biological: Pneumococcal Vaccine, Polyvalent (23-valent) — Administered as an injection at 24 months of age
Biological: Pneumococcal Conjugate Vaccine, Heptavalent — Administered as an injection at 0, 2, 4, and 15 months of age
  Arms: 1
Biological: Placebo — Administered at 0, 2, 4, and 15 months of age
  Arms: 2

SUMMARY:
To assess whether HIV-infected infants who receive a heptavalent pneumococcal conjugate vaccine have more local reactions at the site of injection and systemic reactions than placebo subjects. To assess whether this vaccine is more immunogenic than placebo following the third vaccination.

Children with HIV infection are at increased risk for invasive pneumococcal infection, particularly bacteremia. A large proportion of pneumococcal disease is caused by a limited number of serotypes. The maximum number of pneumococcal serotypes that can be included in a new conjugate vaccine is felt to be limited by the amount of carrier protein. A heptavalent pneumococcal conjugate vaccine has been developed that consists of pneumococcal capsular saccharides from serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F bound to a diphtheria toxin mutant carrier protein.

DETAILED DESCRIPTION:
Children with HIV infection are at increased risk for invasive pneumococcal infection, particularly bacteremia. A large proportion of pneumococcal disease is caused by a limited number of serotypes. The maximum number of pneumococcal serotypes that can be included in a new conjugate vaccine is felt to be limited by the amount of carrier protein. A heptavalent pneumococcal conjugate vaccine has been developed that consists of pneumococcal capsular saccharides from serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F bound to a diphtheria toxin mutant carrier protein.

Infants are randomized to receive either heptavalent pneumococcal conjugate vaccine or placebo by intramuscular injection at study months 0, 2, and 4, and then at 15 months of age. Additionally, patients receive PNU-IMUNE 23 ( pneumococcal polyvalent vaccine ) at 24 months of age.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antipyretics for rectal temperature >= 100.4 F.
* Antiretroviral therapy.

Patients must have:

* HIV positivity.
* Birth weight at least 1800 g (3.75 lb).
* Consent and compliance of parent or guardian.

NOTE:

* Coenrollment in other therapeutic protocols (except ACTG 218, 230, and 279) is permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Enrollment in HIV vaccine trials.
* Major congenital anomalies that are incapacitating, result in immunologic abnormalities, or require major surgical procedures.
* Congenital immunoglobulin deficiency, SS or SC hemoglobinopathy, or asplenia.
* Hypogammaglobulinemia.

Concurrent Medication:

Excluded:

* Prophylactic antipyretics.

Patients with the following prior conditions are excluded:

Acute moderate to severe intercurrent illness or fever within 72 hours prior to study entry.

Prior Medication:

Excluded:

* Any prior pneumococcal vaccine.
* Measles vaccine within 1 month prior to study vaccination.
* Any other routine vaccine within 1 week prior to study vaccination.
* Any immunosuppressant agent, including prednisone, for more than 6 weeks.

Prior Treatment:

Excluded:

* Blood products within 56 days prior to study vaccination.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Comparison of adverse reactions between PCV and placebo patients that occur within 48 hours after each injection | Throughout study
Comparison of seroconversion rates and changes in (IgG) ELISA antibody levels between PCV and placebo patients after the primary series | Throughout study

SECONDARY OUTCOMES:
Comparison of booster rates in serum ELISA (IgG) antibody levels just before the 4th vaccination and one month after the 4th vaccination in children receiving PCV and placebo | Prior to 4th vaccination and at 1 month after 4th vaccination
Comparison of serum IgG1 and IgG2 subclass and IgA type specific seroconversion rates and changes in antibody levels in response to the primary immunization series and booster vaccination between PCV and placebo patients | Throughout study
To compare the decline of serum total IgG, IgG1, IgG2, and IgA pneumococcal type specific antibody after the 3rd and after the 4th vaccination in PCV versus placebo patients | At a time after the 3rd vaccination and at a time after the 4th vaccination
Modeling of the rates of seroconversion and changes in serum antibody levels in PCV patients, after the primary series and booster series, to clinical HIV staging and T-lymphocyte parameters, as well as B-lymphocyte parameters | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: James King, Jr, M.D., Study Chair — University of Maryland, College Park; Sharon Nachman, M.D., Study Chair — SUNY at Stony Brook
Locations (33):
- United States (31):
  - Usc La Nichd Crs, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - San Francisco Gen. Hosp., San Francisco, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - Johns Hopkins Hosp. & Health System - Dept. of Peds., Div. of Infectious Diseases, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - NJ Med. School CRS, Newark, New Jersey
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan